CLINICAL TRIAL: NCT00479726
Title: Lilly's Emotional and Physical Symptoms of Depression Study
Brief Title: Lilly's Emotional and Physical Symptoms of Depression Study (LEAPS)
Acronym: LEAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8300; F1J-MC-HMCY; NCT00479414 (obsolete NCT alias); NCT00479453 (obsolete NCT alias)
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: duloxetine hydrochloride

SUMMARY:
To assess the effectiveness of duloxetine administered once daily in patients with Major Depressive Disorder in a practice based setting

DETAILED DESCRIPTION:
To assess physical and emotional symptoms of depressed patients

ELIGIBILITY:
Inclusion criteria:

* Meet criteria for major depressive disorder according to the DSM-IV diagnostic criteria
* Outpatients at least 18 years of age
* Sign the informed consent
* All females must test negative for a urine pregnancy test at visit 1. Females of child bearing potential must agree to utilize medically acceptable and reliable means of birth control
* Have a level of understanding sufficient to communicate with the investigator and are able to complete all patient self-rated scales in the study

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study or immediate family
* Are employed by Eli Lilly and Company
* Have received treatment within the last 30 days or are currently enrolled in a study with a drug that has not received regulatory approval for any indication at time of study entry
* Current substance dependence, excluding nicotine and caffeine
* Treatment with a monoamine oxidase inhibitor within 14 days prior to visit 1 or potential need to use an MAOI within 5 days after discontinuation of study drug
* Acute liver injury or severe (Child-Pugh Class C) cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 2004-08; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression of Severity
Somatic Symptom Inventory
Depressive Symptomatology-Self Report

SECONDARY OUTCOMES:
Patient Global Impression of Improvement
Mood and Physical Symptoms in Depression
Quality of Life Enjoyment Satisfaction Questionnaire-Short form

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial,contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Wohlreich MM, Wiltse CG, Desaiah D, Ye W, Robinson RL, Kroenke K, Kornstein SG, Greist JH. Duloxetine in practice-based clinical settings: assessing effects on the emotional and physical symptoms of depression in an open-label, multicenter study. Prim Care Companion J Clin Psychiatry. 2007;9(4):271-9. doi: 10.4088/pcc.v09n0404. PMID 17934551
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com